CLINICAL TRIAL: NCT03251144
Title: In Vitro and in Vivo Studies of the Relative Mitochondrial Toxicity of Tenofovir Alafenamide (TAF) vs. Tenofovir Disoproxil Fumarate (TDF)
Brief Title: Relative Mitochondrial Toxicity of Tenofovir Alafenamide (TAF) vs. Tenofovir Disoproxil Fumarate (TDF)
Acronym: UCLACAREMITO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Theodoros Kelesidis, MD, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CO-US-311-4393; CO-US-311-4393 (Other Grant/Funding Number: GILEAD)
Record Dates: First submitted 2017-08-06; First posted 2017-08-16 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: HIV/AIDS; Antiviral Toxicity; Antiviral Drug Adverse Reaction; Mitochondrial Alteration
Keywords: HIV/AIDS; Tenofovir disoproxil fumarate (TDF); Tenofovir alafenamide (TAF); mitochondria; toxicity
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Switch to E/C/FTC/TAF daily (Experimental): Intervention: Participants will be asked to switch antiretrovirals (ART) for a period up to 12 months and mitochondrial physiology will be assessed using a variety of assays. The new ART will be
  1. If the participant is on an ART other than Elvitegravir (ELV)/cobicistat CO)/emtricitabine (FTC)/tenofovir (TDF)] (E/C/FTC/TDF) then the participant will be asked to switch to E/C/FTC/TDF for up to 6 months. This will allow for future switch (after these 6 months) from E/C/FTC/TDF 1 tablet once daily to E/C/FTC/ tenofovir alafenamide (TAF) 1 tablet once daily for a period of 12 months.
  2. If the participant is on E/C/FTC/TDF 1 tablet once daily then the participant will be asked to switch from /C/FTC/TDF 1 tablet once daily to /C/FTC/TAF 1 tablet once daily for a period of 12 months.
  Interventions: Drug: Switch to E/C/FTC/TAF daily

INTERVENTIONS:
Drug: Switch to E/C/FTC/TAF daily — If the participant is on an antiretroviral regimen other than Elvitegravir (ELV)/cobicistat CO)/emtricitabine (FTC)/tenofovir (TDF)] (E/C/FTC/TDF) then the participant will be asked to switch to E/C/FTC/TDF for up to 6 months. This will allow for future switch (after these 6 months) from E/C/FTC/TDF 1 tablet once daily to elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/FTC/TAF) 1 tablet once daily for a period of 12 months.
  b) If the participant is on E/C/FTC/TDF 1 tablet once daily then the participant will be asked to switch from /C/FTC/TDF 1 tablet once daily to /C/FTC/TAF 1 tablet once daily for a period of 12 months.
  Other Names: E/C/FTC/TDF 1 tablet once daily

SUMMARY:
Increased comorbidities such as cardiovascular disease (CVD), are emerging problems in HIV infection but the mechanisms are unclear. Understanding how antiretrovirals can minimize morbidity in treated HIV infection is a research priority. Nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs) are included in all HIV treatment regimens. Tenofovir (TFV) disoproxil fumarate (TDF) has been associated with an increased risk of nephrotoxicity and bone disease compared with other NRTIs. Tenofovir alafenamide (TAF) is an oral prodrug of TFV, but is more stable in plasma as compared with TDF and lower plasma levels of TFV are thought to lead to the favorable safety profile of TAF. Mitochondrial dysfunction has a key role in HIV pathogenesis and may be the common denominator that drives pathogenesis of several comorbidities. Despite the better safety profile of newer (such as TDF) compared to older NRTIs, there are concerns for the potential for longer term toxicity of NRTIs since the exact cellular effects of NRTIs remain unclear. It is unknown whether a four-fold increase in intracellular drug levels seen in peripheral blood mononuclear cells (PBMCs) with TAF may increase toxicity in mitochondria. Better understanding of these effects could provide insights into mechanisms of HIV pathogenesis and selection of NRTIs that improve morbidity in chronic HIV infection.

Hypothesis: Despite higher intracellular levels, TAF has minimal mitochondrial toxicity compared to TDF in vivo. This research will explore the relative mitochondrial toxicity of newer NRTIs (TAF, TDF) as a possible mechanism for differential NTRI-related toxicities. These data will allow selection of NRTIs that may improve morbidity in chronic treated HIV infection. Towards this aim, the investigators will use a robust experimental approach to study NRTI-related mitochondrial dysfunction using novel methods, human cell lines and PBMC. Our specific aims are: Aim 1: To evaluate the relative in vitro effects of TAF and TDF compared to an older NRTI (ddC) on 5 independent measures of mitochondrial function in the human cell line HepG2 and PBMC. Aim 2: To explore in vivo whether there is increased mitochondrial dysfunction with the use of TAF vs. TDF in chronic treated HIV infection. The investigators anticipate that the proposed experimental approach will set the basis for future large scale studies to directly compare subtle potential mitochondrial toxicities of newer NRTIs in large HIV cohorts.

DETAILED DESCRIPTION:
Increased comorbidities such as cardiovascular disease (CVD), bone and kidney disease are emerging problems in HIV infection but the mechanisms are unclear. Understanding how antiretrovirals can minimize morbidity in treated HIV infection is a research priority. Nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs) are included in all HIV treatment regimens. Tenofovir (TFV) disoproxil fumarate (TDF) has been associated with an increased risk of nephrotoxicity and bone disease compared with other NRTIs. Tenofovir alafenamide (TAF) is an oral prodrug of TFV, but is much more stable in plasma as compared with TDF and markedly lower plasma levels of TFV are thought to lead to the favorable safety profile of TAF. Mitochondrial dysfunction has a key role in HIV pathogenesis and may be the common denominator that drives pathogenesis of several comorbidities. Despite the better safety profile of newer (such as TDF) compared to older NRTIs, there remain concerns for the potential for longer term toxicity of the current NRTIs especially since the exact cellular effects of NRTIs remain unclear. It is unknown whether a four-fold increase in intracellular drug levels seen in peripheral blood mononuclear cells (PBMCs) with TAF may increase toxicity in mitochondria. Better understanding of these effects could provide insights into mechanisms of HIV pathogenesis and selection of NRTIs that improve morbidity in chronic HIV infection.

Hypothesis: Despite higher intracellular levels, TAF has minimal/no overall mitochondrial toxicity compared to TDF in vivo. The investigators anticipate that the preliminary data and the proposed experimental approach will set the basis for future large scale studies to directly compare subtle potential mitochondrial toxicities of newer NRTIs in large HIV cohorts.

Primary Objective: This research application will explore the relative mitochondrial toxicity of newer NRTIs (TAF, TDF) as a possible mechanism for differential NTRI-related toxicities. These data will allow selection of NRTIs that may improve morbidity in chronic treated HIV infection, given the known possible role of mitochondrial dysfunction in pathogenesis of HIV-related comorbidities. Towards this aim, the investigators will use a robust experimental approach to study NRTI-related mitochondrial dysfunction using novel methods, human cell lines and PBMC. The specific aims of this project are: Aim 1: To evaluate the relative in vitro effects of TAF and TDF compared to an older NRTI (ddC) on 5 independent measures of mitochondrial function in the human cell line HepG2 and PBMC. Hypothesis: Despite higher intracellular levels, TAF has minimal/no overall mitochondrial toxicity compared to TDF in both the HepG2 line and PBMC. ddC will be used as a positive control for NRTI-induced mitochondrial dysfunction. Aim 2: To explore in vivo whether there is increased mitochondrial dysfunction with the use of TAF vs. TDF in chronic treated HIV infection. The overall goal of this proposal is to determine the in vitro and in vivo effects of TAF on mitochondria.

Treatment regimen: Healthy HIV-uninfected > 18 years old with no known comorbidities including metabolic disease will be recruited for PBMC isolation for the in vitro studies described in Aim 1 (n=30). For Aim 1, cells will be exposed to 10 μM (and other dose that will be determined after discussions with Gilead) NRTIs (TDF, TAF, ddC) for up to 14 days of treatment. To evaluate the relative mitochondrial toxicity of TDF vs. TAF in vivo (Aim 2), an open-label switch study will be conducted in virologically-suppressed, HIV-1 positive participants. The switch regimen will be Stribild® (elvitegravir 150 mg/cobicistat 150 mg/emtricitabine 200 mg/tenofovir disoproxil fumarate 300 mg; E/C/F/TDF) to Genvoya® (elvitegravir 150 mg/cobicistat 150 mg/emtricitabine 200 mg/tenofovir alafenamide 10 mg; E/C/F/TAF). For inclusion and exclusion criteria see respective sections.

Primary Endpoint: Overall, the above in vitro and in vivo measurements of mitochondrial function before and after TAF and TDF will test the hypotheses that newer NRTIs have minimal overall mitochondrial toxicity in humans. From all the measures of mitochondrial function, cellular oxygen consumption (COC; as determined by Seahorse technology) will be considered the "gold standard" given it is a measure of the most important mitochondrial function (oxidative phosphorylation) that relates to clinical outcome. Given the uncertainty of what measure of mitochondrial function can best predict NRTI-induced mitochondrial toxicity, comparison of relative fold induction of mitochondrial dysfunction in PBMC vs. HepG2 cells in response to a specific concentration of a known NRTI inducer of mitochondrial dysfunction (ddC) will be used to guide analysis. The baseline measurement will be used to control for confounders of NRTI-related mitochondrial dysfunction (each person will serve as his/her own control) and results will be expressed as relative-fold change compared to baseline. In addition, using similar approach, Aim 2 will explore whether switch from TDF to a TAF-based regimen will induce any changes in measures of mitochondrial function. This approach ensures that any changes in the mitochondrial function at 6 and/or 12 months will be secondary only to the NRTI switch.

Secondary Endpoints: It is accepted that two independent measures of mitochondrial function can more reliably predict mitochondrial dysfunction compared to each one of the measures separately. The investigators will define NRTI-induced mitochondrial toxicity as significant change in any of other major measures of mitochondrial toxicity [reduction in membrane potential (Δψm), increase in mitochondrial reactive oxygen species (mito-ROS), decrease in the amount of mitochondrial DNA (mtDNA), abnormal mitochondrial dynamics (increase fragmentation of mitochondria)). Finally, other exploratory secondary endpoints (based on available left-over resources) will be measurement of intracellular levels of TAF metabolites. Flow cytometry and live cell imaging will be determined as needed.

The investigators will define NRTI-induced mitochondrial toxicity as significant change in any of the measures of mitochondrial toxicity (COC, Δψm, mito-ROS, mtDNA, mitochondrial dynamics). The baseline measurement will be used to control for confounders of NRTI-related mitochondrial dysfunction (each person will serve as his/her own control) and results will be expressed as relative-fold change compared to baseline. In addition, using similar approach, Aim 2 will explore whether switch from TDF to a TAF-based regimen will induce any changes in measures of mitochondrial function. This approach ensures that any changes in the mitochondrial function at 6 and/or 12 months will be secondary only to the NRTI switch.

Since each donor will contribute samples to all experimental groups (baseline, follow up measurement), paired t-test, linear mixed effects model and nonparametric test (as needed) will be used to compare expression measures between groups adjusting for donor effects (age, sex, race.

The results from this research will yield useful information on NRTI-related overall mitochondrial dysfunction that can further be validated in large studies with data on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for HIV negative participants

All HIV negative participants must meet the following criteria:

1. 18 years of age or older
2. Understands and agrees to local STI reporting requirements
3. HIV negative at screening by self-report, with no significant medical diagnoses
4. HIV negative by both HIV antibody and HIV PCR in blood (samples obtained during Visit 1)
5. Able and willing to communicate in English
6. Able and willing to provide written informed consent to take part in the study
7. Able and willing to provide adequate information for locator purposes
8. Able and willing to provide medical/surgical history
9. Availability to return for all study visits, barring unforeseen circumstances
10. Willing to abstain from insertion of anything (drug, enema, penis or sex toy) in rectum for 12 hours before and 72 hours after each flexible sigmoidoscopy

    In addition to the criteria listed above, female participants must meet the following criteria
11. Negative pregnancy test
12. Post-menopausal or using and acceptable form of contraception (e.g. barrier method, IUD, hormonal contraception, or surgical sterilization).

HIV participant inclusion criteria

Specific enrollment inclusion criteria include:

* 18 years of age or older
* Cases: Chronically infected and on anti-retroviral therapy with suppressed viremia (viral RNA <50 copies per ml)
* On stable antiretroviral therapy for 6 months with either a) Stribild®; elvitegravir 150 mg/cobicistat 150 mg/emtricitabine 200 mg/tenofovir disoproxil fumarate 300 mg; E/C/F/TDF)
* Adequate renal function determined by the Cockcroft-Gault formula for creatinine clearance (>60 mL/min/1.73 m2
* Controls: HIV negative as documented in prior tests and willing to undergo repeat HIV testing
* Able and willing to communicate in English
* Able and willing to provide written informed consent to take part in the study

Exclusion Criteria:

* Exclusion criteria for all study participants:

Participants who meet any of the following criteria at screening will be excluded from the study:

1. History of chronic inflammatory bowel disease, radiation proctitis or other chronic gastrointestinal disease, exclusive of functional bowel disease (irritable bowel syndrome)
2. History of significant gastrointestinal bleeding
3. History of a bleeding disorder
4. History of colostomy
5. History of auto-immune diseases
6. Chronic viral hepatitis
7. History of diabetes
8. History of chemotherapy (for cancer or organ transplantation)
9. The chronic or recent (~2 weeks) use of antimitotic drugs, sulfonamides or antibiotics
10. History of or current coagulopathy and/or on anticoagulant therapy
11. Anticipated use or unwillingness to abstain from use of aspirin, NSAIDS or any other drugs (including over the counter products) that are associated with the increased likelihood of bleeding
12. Active rectal infection (gonorrhea, chlamydia trachomatis, or HSV)
13. Positive STI at screening (urine NAAT)

    o Participants will be allowed one re-screening visit after appropriate STI treatment
14. History of underlying cardiac arrhythmia or renal disease
15. History of severe recent cardiac or pulmonary event
16. > Grade 2 laboratory abnormality at baseline that can not be documented as stable /chronic for that individual
17. Any other condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological or cerebral disease.
18. Pregnancy
19. Breastfeeding
20. Female of child-bearing potential unwilling to use acceptable form of contraception

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodoros Kelesidis, MD, PhD, Msc, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA CARE Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Assignment based on inclusion criteria TAF based vs TDF based antivirals
Groups:
- TAF Based ART: HIV infected persons who receive TAF based ART
- TDF Based ART: HIV infected persons who receive TDF based ART
Period: Overall Study
Arm/Group | TAF Based ART | TDF Based ART
Started | 15 | 11
Completed | 15 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients on TAF based vs TDF based ART
Groups:
- Total: Total of all reporting groups
Arm/Group | TAF Based ART | TDF Based ART | Total
Number analyzed (Participants) | 15 | 11 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 11 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 11 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 13 | 9 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Mitochondrial Function [Cellular Oxygen Consumption (COC)] Over 12 Months After Switch of Antiretrovirals.
Description: Change in mitochondrial function [abnormal mitochondrial dynamics [(cellular oxygen consumption (COC)] over 12 months after switch of antiretrovirals.
Time Frame: 12 month visit after switch
Measure: Median (Inter-Quartile Range); unit: pmoles O2/min
Arm/Group | TAF Based ART | TDF Based ART
Number analyzed (Participants) | 15 | 11
pmoles O2/min | 50 [42 to 58] | 70 [65 to 72]
Statistical Analysis 1: Comparison: TAF Based ART vs TDF Based ART; Test type: Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 20, Standard Error of Mean 3.0

ADVERSE EVENTS:
Time Frame: Up to 9 months
Arm/Group | TAF Based ART | TDF Based ART
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/11
Other Adverse Events (participants affected / at risk) | 0/15 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT03251144/Prot_SAP_000.pdf